CLINICAL TRIAL: NCT06550830
Title: A Randomized, Double-blind, Controlled Combined With Open-label Phase Ia Clinical Trial to Evaluate the Safety and Immunogenicity of 24-valent Pneumococcal Conjugate Vaccine in Children Aged 2-17 Years.
Brief Title: Clinical Trial of PCV24 in Children Aged 2-17 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV24-1002
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple for children aged 2-5 years; open-label for children aged 6-17 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): 12 participants aged 6-17 years and 30 participants aged 2-5 years will be randomized to receive Sinovac PCV24 formulation 1. Route of administration is intramuscular injection at deltoid muscle of upper arm.
  Immunization schedule is 1 dose.
  Interventions: Biological: Sinovac PCV24 formulation 1
- Experimental group 2 (Experimental): 12 participants aged 6-17 years and 30 participants aged 2-5 years will be randomized to receive Sinovac PCV24 formulation 2. Route of administration is intramuscular injection at deltoid muscle of upper arm.
  Immunization schedule is 1 dose.
  Interventions: Biological: Sinovac PCV24 formulation 2
- Active control group (Active Comparator): 30 participants aged 2-5 years will be randomized to receive Prevenar13®. Route of administration is intramuscular injection at deltoid muscle of upper arm.
  Immunization schedule is 1 dose.
  Interventions: Biological: Prevenar13®

INTERVENTIONS:
Biological: Sinovac PCV24 formulation 1 — One dose of Sinovac PCV24 formulation 1(0.5mL)
  Arms: Experimental group 1
Biological: Sinovac PCV24 formulation 2 — One dose of Sinovac PCV24 formulation 2(0.5mL)
  Arms: Experimental group 2
Biological: Prevenar13® — One dose of PCV13 manufactured by Pfizer
  Arms: Active control group

SUMMARY:
A Phase Ia clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Sinovac Life Science Co., Ltd will be conducted in children aged 2-17 years. The objective of the study is to evaluate the safety and immunogenicity of Sinovac PCV24. The trial is a randomized, double-blind, controlled combined with open-label phase Ia clinical trial.

DETAILED DESCRIPTION:
A phase Ia clinical trial of the study of 24-valent Pneumococcal Conjugate Vaccine (PCV24) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in Chinese children aged 2-17 years. The trial is a randomized, double-blind, controlled combined with open-label study. The objective of this study is to evaluate the safety and immunogenicity of PCV24 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine for participants aged 2-5 years is the Prevenar13® manufactured by Pfizer.

A total of at least 114 participants will be enrolled, including 24 children aged 6-17 years and 90 children aged 2-5 years. Children aged 6-17 years will receive PCV24 formulation 1 and PCV24 formulation 2 in a 1:1 ratio. Children aged 2-5 years will receive PCV24 formulation 1, PCV24 formulation 2 and Prevenar13® in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who are aged 2-17 years;
2. Participants and their guardians provide legal proof of identity, as well as vaccination record (for children aged 2-5 years);
3. Participants' guardians understand and voluntarily sign the informed consent form; participants aged 8-17 years sign the written assent;
4. Participants can follow all study procedures and stay in contact during the study.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment;
2. History of invasive pneumococcal diseases (IPDs) or other pneumococcal diseases caused by Streptococcus pneumoniae, as confirmed by laboratory tests;
3. History of allergy or adverse reactions to the vaccine or vaccine components, or history of allergy, such as urticaria, dyspnea, angioedema and anaphylactic shock;
4. Congenital malformations or developmental disorders, genetic defects (such as Down syndrome, thalassemia, or G6PD deficiency), severe malnutrition;
5. Have uncontrolled chronic diseases or history of severe diseases, including but not limited to cardiovascular diseases, such as cardiovascular diseases (e.g. congenital heart disease), metabolic diseases (such as diabetes), hematological diseases (e.g. severe anemia),liver and kidney diseases, digestive diseases, respiratory diseases (such as active tuberculosis), malignant tumors and major functional organ transplantation history;
6. Autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection)
7. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets level), history of obvious bleeding, hematoma or bruising after intramuscular injection or venipuncture.
8. Have/have suffered from a serious neurological disorder (epilepsy or convulsions) or mental illness or have a family history of such diseases.
9. Long-term alcohol or drug abuse.
10. Have received > 14 days of immunosuppressive or other immunomodulatory therapy in the past 6 months, or cytotoxic therapy, or plan to receive such therapy during the study period.
11. Received immunoglobulin or other blood products within 3 months prior to enrollment, or plan to receive such treatment during the study period;
12. Received other investigational drugs or vaccines within 30 days prior to enrollment, or plan to receive such drugs or vaccines during the study;
13. Received live attenuated vaccine within 14 days prior to enrollment;
14. Received subunit or inactivated or other vaccine within 7 days prior to enrollment;
15. Acute diseases or acute onset of chronic diseases within 7 days prior to enrollment, or known or suspected active infection;
16. Women who are pregnant or breastfeeding (if applicable);
17. Abnormalities in clinical laboratory indicators that exceed reference range and are clinically significant.
18. Had fever (axillary temperature> 37.0℃) before vaccination;
19. In the investigator's judgment, the participant has any other factors that make him or her unfit to participate in the clinical trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 0-30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions | 0-7 days after vaccination
  Incidence of adverse reactions within 7 days after vaccination
Incidence of serious adverse events (SAE) | 0-6 months after vaccination
  Incidence of SAE during the period of safety monitoring
Incidence of clinically significant abnormality in laboratory examination tests | 0-3 days after vaccination
  Incidence of clinically significant abnormality in blood routine, blood biochemistry and urine routine test results within 3 days after vaccination
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after vaccination
  IgG GMC 30 days after vaccination
Proportion of Pneumococcal serotype-specific IgG antibody concentration ≥0.35 μg/ml (seropositive rate) | 30 days after vaccination
  Proportion of IgG antibody concentration ≥0.35 μg/ml
Proportion of Pneumococcal serotype-specific IgG antibody concentration ≥1.0 μg/ml | 30 days after vaccination
  Proportion of IgG antibody concentration ≥1.0 μg/ml
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after vaccination
  IgG GMI 30 days after vaccination
Proportion of pneumococcal serotype-specific IgG antibody concentration increase≥4 | 30 days after vaccination
  Proportion of IgG antibody concentration increase≥four folds 30 days after vaccination
Pneumococcal serotype-specific opsonophagocytic assay (OPA) geometric mean titer (GMTs) | 30 days after vaccination
  OPA GMT 30 days after vaccination
Pneumococcal serotype-specific OPA GMI | 30 days after vaccination
  OPA GMI 30 days after vaccination
Proportion of Pneumococcal serotype-specific OPA GMT≥1:8 | 30 days after vaccination
  Proportion of Pneumococcal serotype-specific OPA GMT≥1:8 30 days after vaccination
Proportion of pneumococcal serotype-specific OPA antibody titer increase≥4 | 30 days after vaccination
  Proportion of OPA antibody titer increase≥four folds 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kai Chu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention (Jiangsu Provincial Academy of Preventive Medicine)
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention (Jiangsu Provincial Academy of Preventive Medicine), Nanjing, Jiangsu, China